CLINICAL TRIAL: NCT03249467
Title: Validation of the French Version of the Health Assessment Questionnaire II (HAQ-II) for Rheumatoid Arthritis
Acronym: HAQ-II
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3030_HAQ-II
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
Keywords: HAQ-II; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to develop a validated French version of the HAQ-II questionnaire for rheumatoid arthritis.

DETAILED DESCRIPTION:
The HAQ is the original Health Assessment Questionnaire used in rheumatology. It is available in more than 60 languages and includes 42 items. However the questionnaire is not easy to use in the clinic : complicated questions, long to answer for the patient and not easy to score for the doctor.

The HAQ-II is a reliable and valid 10-item questionnaire that performs at least as well as the HAQ and is simpler to administer and score. It includes 5 items already translated in English and 5 new items not yet translated.

The aim of the study is the validation of the French version of the HAQ-II for rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient with rheumatoid arthritis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-10-17 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Internal validity, scale HAQ-II | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France